CLINICAL TRIAL: NCT05583474
Title: A Phase III, Multi-center, Randomized, Single-blind (to Evaluator), Parallel, and Positive-controlled Clinical Trial Evaluating the Efficacy and Safety of OPC-1085EL Ophthalmic Solution in the Treatment of Primary Open Angle Glaucoma or Ocular Hypertension in Chinese Subjects
Brief Title: OPC-1085EL in the Treatment of Primary Open Angle Glaucoma or Ocular Hypertension in Chinese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001-403-00013
Record Dates: First submitted 2022-10-08; First posted 2022-10-17 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Open Angle Glaucoma or Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subject receive OPC-1085EL solution (Experimental): OPC-1085EL group ，one drop for each eye, once per day for 8 weeks
  Interventions: Drug: OPC-1085EL
- subject receive 0.005% latanoprost ophthalmic solution (Active Comparator): 0.005% latanoprost ophthalmic solution group ，one drop for each eye, once per day for 8 weeks
  Interventions: Drug: 0.005% Latanoprost

INTERVENTIONS:
Drug: OPC-1085EL — one drop for each eye, once per day
  Other Names: OPC-1085EL ophthalmic solution
  Arms: subject receive OPC-1085EL solution
Drug: 0.005% Latanoprost — one drop for each eye, once per day
  Other Names: 0.005% Latanoprost ophthalmic solution
  Arms: subject receive 0.005% latanoprost ophthalmic solution

SUMMARY:
It is a phase III, multi-center, randomized, single-blind (to evaluator), parallel, and positive-controlled clinical trial evaluating the efficacy and safety of OPC-1085EL in the treatment of primary open angle glaucoma or ocular hypertension in Chinese subjects. It is planned that 240 subjects (120 in each group) will be randomly assigned to receive OPC-1085EL or 0.005% latanoprost ophthalmic solution (latanoprost) at a ratio of 1:1.

DETAILED DESCRIPTION:
The trial includes 2 period:

1. Screening period: 4 weeks. For subjects entering the screening period, 0.005% latanoprost will be administered for 4 consecutive weeks, one drop for each eye, once per day.
2. Evaluation period: 8 weeks. Subjects who are eligible are randomly assigned to the OPC-1085EL group or 0.005% latanoprost group at a ratio of 1:1, one drop for each eye, once per day.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Unlimited
2. Hospitalization status: Outpatients
3. Age: 20-80 years old
4. Subjects with both eyes diagnosed as primary open angle glaucoma or ocular hypertension.

   [At the end of the screening period]
5. IOP: After 4 weeks treatment with 0.005% latanoprost, the unilateral eye with a pre-dose IOP from 18 mmHg to <30 mmHg, and IOP <30 mmHg in the contralateral eye.

Exclusion Criteria:

1. Subjects with a best-corrected visual acuity ≤ 0.2.
2. Subject with any secondary glaucoma such as exfoliative or pigmented glaucoma.
3. Subjects who cannot stop using contact lenses during the trial.
4. Subjects who are judged by investigators to be at risk when receiving carteolol hydrochloride or 0.005% latanoprost as monotherapy.
5. Subjects who are allergic to any ingredients in carteolol or latanoprost.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
evaluate pre-dose intraocular pressure change from baseline to week 8 | baseline；week 8
  Baseline intraocular pressure: The pre-dose and 2 hours after dosing intraocular pressures measured

SECONDARY OUTCOMES:
intraocular pressure | Week 4；Week 8:
  evaluate the effects of OPC-1085ELv.s.0.005% latanoprost by measure intraocular pressure
intraocular pressure change from baseline | Week 4；Week 8
  evaluate the effects of OPC-1085ELv.s.0.005% latanoprost by measure intraocular pressure
intraocular pressure change rate from baseline | week 4:
  intraocular pressure change rate=(intraocular pressure change from baseline at each time point)/ (corresponding baseline intraocular pressure) × 100%
Safety evaluation variable：adverse event | from screening period to evaluation period, assessed up to 3 weeks.
  adverse event start date, end date, seriousness, severity, relationship to trial treatment (IMP causality), action taken with trial treatment, and outcome will be collect.

CONTACTS AND LOCATIONS:
Overall Officials: Huaixing Sun, Doctor, Principal Investigator — Eye & ENT Hospital of Fudan University
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No